CLINICAL TRIAL: NCT06332287
Title: A Prospective, Single-arm, and Exploratory Phase II Clinical Study of Trilaciclib Combined With Lateral Ventricular Chemotherapy in the Treatment of Advanced Non-small Cell Lung Cancer With Leptomeningeal Metastasis
Brief Title: A Study of Trilaciclib Combined With Chemotherapy in the Treatment of Advanced NSCLC With Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-NSCLC
Record Dates: First submitted 2024-03-12; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Intervention Model Description: Trilaciclib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib+Pemetrexed (Experimental): Patients were treated with Trilaciclib (240mg/m2, administered within 4 hours before each chemotherapy,Q3W) and pemetrexed (30mg,Q3W) until disease progression as assessed by the investigator according to RECIST 1.1 criteria or withdrawal or discontinuation criteria were met.
  Interventions: Drug: combination of Trilaciclib and Pemetrexed

INTERVENTIONS:
Drug: combination of Trilaciclib and Pemetrexed — This was a single-arm, exploratory study of the combination of Trilaciclib and Pemetrexed in patients with non-small cell lung cancer with leptomeningeal metastasis. Observed the incidence of chemotherapy-induced myelosuppression, and imaging was performed every six cycles to assess tumor response.
  Other Names: G1T28; CDK 4/6 inhibitor

SUMMARY:
To observe the efficacy of Trilaciclib combined with lateral ventricular chemotherapy in the treatment of non-small cell lung cancer with leptomeningeal metastasis。

DETAILED DESCRIPTION:
A single-arm, open-label, interventional study was conducted in 25 NSCLC patients with leptomeningeal metastases to observe the efficacy of Trilaciclib combined with lateral ventricular chemotherapy in the treatment of non-small cell lung cancer with leptomeningeal metastases, and to evaluate the incidence and duration of severe neutropenia in the first cycle.

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years when fisrt dose of Trilaciclib, regardless of gender；
* ECOG-PS score of 0-1，and no worsening in the 2 weeks before the study drug；
* expected survival≥12 weeks；
* Advanced non-small cell lung cancer with leptomeningeal metastasis；
* with an Ommaya sac has been implanted；
* At least one measurable lesion meeting RECIST1.1 criteria was present；
* Laboratory tests met the following criteria: hemoglobin ≥100 g/L (female), 110g/L (male) ；neutrophil count ≥ 2×109/L ；platelet count ≥100×109/L; Creatinine ≤ 15mg/L or creatinine clearance (CrCl) ≥ 60 mL/min (Cockcroft-Gault formula); Total bilirubin ≤ 1.5× upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN or 5× ULN (for patients with liver metastases); Albumin ≥ 30 g/L;
* Patients of reproductive age(including female and male patients'female companions)must use effective birth control measures;
* Voluntarily participate and sign informed consent;

Exclusion Criteria:

* Patients of reproductive age(including female and male patients'female companions)must use effective birth control measures;
* Stroke or cardio-cerebrovascular event within 6 months before enrollment;
* QTcF interval > 480msec at screening, QTcF > 500msec for patients with implanted ventricular pacemakers;
* Previous hematopoietic stem cell or bone marrow transplantation;
* Allergy to the study drug or its components;
* If the investigator considers that it is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Duration of severe neutropenia (DSN) | During Trilaciclib plus chemotherapy assessed up to 21 days
  Duration of severe neutropenia in cycle 1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  Occurrence and severity of AEs by NCI CTCAE v5.0
Incidence of grade 3 and 4 hematologic toxicity | during Trilaciclib plus chemotherapy assessed up to 1 years
  Incidence of grade 3 and 4 hematologic toxicity
Incidence of G-CSF treatment | during Trilaciclib plus chemotherapy assessed up to 1 years
  Incidence of G-CSF treatment
Incidence of platelet transfusion | during Trilaciclib plus chemotherapy assessed up to 1 years
  Incidence of platelet transfusion

CONTACTS AND LOCATIONS:
Overall Officials: fang S cun, M.D., Study Director — Nanjing Brain Hospital
Locations (1):
- Fang Shencun, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No